CLINICAL TRIAL: NCT06290336
Title: Effect of Prehabilitation Before Total Knee Replacement on Post-operative Patient-reported Joint Awareness, Enablement and Knee Function
Brief Title: Pre-Operative Exercise Therapy and Patient Education Before Total Knee Replacement
Acronym: PROTEKT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Region Östergötland (Other); Region Jönköping County (Other Government)
Responsible Party: Principal Investigator, Joanna Kvist, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROTEKT
Record Dates: First submitted 2024-02-22; First posted 2024-03-04 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis
Keywords: Knee replacement; Exercise therapy; Education; Knee function; Satisfaction
MeSH Terms: conditions — Osteoarthritis, Knee; Personal Satisfaction | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Multi-center randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor blinded to group allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Pre-operative exercise therapy and education before knee replacement surgery
  Interventions: Other: Pre-operative exercise therapy and education; Other: Standardized pre-operative information session
- Control group (Other): Standard care
  Interventions: Other: Standardized pre-operative information session

INTERVENTIONS:
Other: Pre-operative exercise therapy and education — Pre-operative supervised exercise therapy consisting of individualized strength, mobility and balance exercises and continuous education through individual discussions of expectations of post-operative recovery, pain and swelling, course of rehabilitation, long term function and activity level etc. Twice a week, approximately one hour/session.
  Arms: Intervention group
Other: Standardized pre-operative information session — As part of the standard care procedure, patients in the intervention and control group will participate in a standardized pre-operative information session approximately 2 weeks before surgery. General information regarding preparations before surgery (e.g. preparing the home environment), events during the hospital stay and the rehabilitation process after discharge will be provided.

SUMMARY:
The goal of this multi-center randomized controlled trial is to investigate the effect of pre-operative exercise therapy and education for patients awaiting knee replacement surgery on subjective knee function, patient satisfaction and enablement compared to standard care.

The main questions it aims to answer are:

* Does pre-operative exercise therapy and education lead to better subjective knee function compared to standard care one year after surgery?
* Does pre-operative exercise therapy and education lead to a higher level of patient satisfaction compared to standard care one year after surgery?
* Does pre-operative exercise therapy and education lead to better patient enablement compared to standard care six weeks after surgery?
* Does pre-operative exercise therapy and education lead to better objective knee function compared to standard care six weeks after surgery?

Participants will be randomized stratified by age (≤ 67 years, > 67 years) to either pre-operative supervised individualized exercise therapy combined with education two sessions/week (intervention group) or to standard care (control group). The intervention will be continuously ongoing for at least eight weeks from the point of decision for surgery until as close to the surgery as possible.

DETAILED DESCRIPTION:
Eligible patients will be randomized through opaque concealed envelopes stratified by age (≤ 67 years, > 67 years) with a 1:1 allocation ratio into the intervention or the control group, after getting a decision for surgery from the surgeon. Inclusion and exclusion criteria are described in a section below. The envelopes and allocation list will be kept in a locked fire-proof storage in a different building than where the allocation process will take place.

The patients in the intervention group will participate in pre-operative supervised exercise therapy and education, continuously ongoing from point of surgery decision until surgery. Twice a week, approximately one hour/session. Training consists of individualized strength, balance and mobility exercises, and education consists of ongoing individualized discussion regarding patients' expectations of post-operative recovery, pain and swelling, course of rehabilitation, long term function and activity level etc.

Patients in both groups will participate in a standardized pre-operative information session, approximately 2 weeks before surgery. General information regarding preparations before surgery (e.g. preparing the home environment), events during the hospital stay and the rehabilitation process after discharge will be provided as part of the standard care procedure.

Patients in the control group will participate in the standardized pre-operative information session mentioned above. They will not receive any specific information regarding training and exercise or individualized education outside of regular discussion with the surgeon when consenting to/making the decision for surgery.

Baseline and follow-up measures after 8 weeks, 1-2 weeks before surgery and 6 weeks after surgery will include objective and patient reported outcome measures. Follow-up measures 3 months and 1 year after surgery will consist of patient reported outcome measures only.

ELIGIBILITY:
Inclusion Criteria:

* Waiting list for primary unilateral knee replacement surgery
* Osteoarthritis of the knee being the primary reason for surgery
* Reside within 60 minutes of travel to the site of the intervention

Exclusion Criteria:

* Previous knee replacement surgery in the other knee
* Other reason than osteoarthritis of the knee as the primary reason for surgery
* Impaired cognitive function
* Not being independent speaking and reading in swedish language
* Chronic illness or disability etc hindering full participation in the intervention

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Forgotten Joint Score-12 (FJS-12) from baseline to 1 year after surgery | Baseline; 1 year after surgery
  Patient-reported outcome measure (PROM) where patients assesses how aware they are of their affected knee on a 5 item Likert scale in 12 different situations in daily living. The result is summarized into a total result on a 0-100 scale, with 0 being worst (high awareness) and 100 being best (low awareness)
Change in modified Patient Enablement Instrument-2 (Mod-PEI-2) from baseline to 6 weeks after surgery | Baseline; 6 weeks after surgery
  6-item PROM where patients are asked to assess their ability to cope with life, understand and cope with their disease, ability to stay healthy and help themselves etc during the last 4 weeks. Items are answered in a 5-item Likert scale ranging from extremely well to not at all. Results are summarized into a total score from 6 to 30, with higher scores indicating better enablement.

SECONDARY OUTCOMES:
Patient satisfaction at 1 year after surgery | 1 year after surgery
  5 item Likert scale ranging from very dissatisfied to very satisfied
Change in maximal isometric knee extension in 90 degrees of flexion from baseline to 8 weeks after start of intervention and 1-2 weeks before surgery | Baseline; 8 weeks after randomization/start of intervention; 1-2 weeks before surgery
  Seated, using fixed dynamometer
Change in active knee range of motion from baseline to 8 weeks after start of intervention and 1-2 weeks before surgery | Baseline; 8 weeks after randomization/start of intervention; 1-2 weeks before surgery
  Supine, using goniometer
Change in 30sCST from baseline to 8 weeks after start of intervention and 1-2 weeks before surgery | Baseline; 8 weeks after randomization/start of intervention; 1-2 weeks before surgery
  Maximal number of completed repetitions in 30 seconds
Change in Knee Osteoarthritis Outcome Score (KOOS) from baseline to 8 weeks after start of intervention, 1-2 weeks before surgery, 6 weeks, 3 months and 1 year after surgery | Baseline; 8 weeks after randomization/start of intervention; 1-2 weeks before surgery; 6 weeks after surgery; 3 months after surgery; 1 year after surgery
  PROM with 5 sub-categories on different topics regarding pain, symptoms, activities in daily living, sports and recreation and quality of life. Results are summarized in a 0-100 scale with 0 being worst and 100 best
Change in 30 seconds Chair to Stand-Test (30sCST) from baseline to 6 weeks after surgery | Baseline; 6 weeks after surgery
  Maximal number of completed repetitions in 30 seconds
Change in active knee range of motion from baseline to 6 weeks after surgery | Baseline; 6 weeks after surgery
  Supine, using goniometer
Change in maximal isometric knee extension in 90 degrees of flexion from baseline to 6 weeks after surgery | Baseline; 6 weeks after surgery
  Seated, using fixed dynamometer
: Change in EuroQol 5 Dimensions 3 Levels (EQ5D-3L) from baseline to 8 weeks after start of intervention, 1-2 weeks before surgery, 6 weeks, 3 months and 1 year after surgery | Baseline; 8 weeks after randomization/start of intervention; 1-2 weeks before surgery; 6 weeks after surgery; 3 months after surgery; 1 year after surgery
  PROM in five dimensions on different topics of state of health answered in a three-level scale. Values are anchored at 1 (full health) and 0 (a state as bad as being dead), allowing also negative values. The outcome also includes a grading of the patients' perceived state of health on a Visual Analogue Scale (VAS) 0-100, with 0 being worst possible state of health and 100 being best possible state of health
Change in International Physical Activity Questionnaire - short form (IPAQ-sf) from baseline to 8 weeks after start of intervention, 1-2 weeks before surgery, 6 weeks, 3 months and 1 year after surgery | Baseline; 8 weeks after randomization/start of intervention; 1-2 weeks before surgery; 6 weeks after surgery; 3 months after surgery; 1 year after surgery
  PROM in 4 sub-categories with follow-up questions where patients assess their physical activity habits. Results are summarized into three categories; low, moderate or high physical activity
Change in Mod-PEI-2 from baseline to 8 weeks after start of intervention, 1-2 weeks before surgery, 6 weeks, 3 months and 1 year after surgery | Baseline; 8 weeks after randomization/start of intervention; 1-2 weeks before surgery; 3 months after surgery; 1 year after surgery
  6-item PROM where patients are asked to assess their ability to cope with life, understand and cope with their disease, ability to stay healthy and help themselves etc during the last 4 weeks. Items are answered in a 5-item Likert scale ranging from extremely well to not at all. Results are summarized into a total score from 6 to 30, with higher scores indicating better enablement.
Change in FJS-12 from baseline to 8 weeks after start of intervention, 1-2 weeks before surgery and 6 weeks and 3 months after surgery | Baseline; 8 weeks after randomization/start of intervention; 1-2 weeks before surgery; 6 weeks after surgery; 3 months after surgery
  PROM where patients assess how aware they are of their affected knee on a 5 item Likert scale in 12 different situations in daily living. The result is summarized into a total result on a 0-100 scale, with 0 being worst (high awareness) and 100 being best (low awareness)
Change in objectively measured physical activity and sedentary habits via accelerometer, from baseline to 8 weeks after start of intervention, 3 months and 1 year after surgery | Baseline; 8 weeks after randomization/start of intervention; 3 months after surgery; 1 year after surgery
  Physical activity and sedentary habits is objectively measured via the activPAL™ accelerometer. It is attached to the front of the thigh of the affected leg and is worn 24 hours a day for 7 days.

OTHER OUTCOMES:
Adherence | From initiation of the intervention until the 8 week follow-up, and then continuously ongoing if surgery date is schedueled after the 8 week follow up.
  Adherence to the intervention, exercise therapy protocol and education conversations is registered at each session. An exercise journal is kept for all patients and the number of exercises, exercise variations performed, dosage and load used and education topics discussed is recorded.
Description of surgical procedures | 6 weeks after surgery
  Information about surgical procedure specifics, such as type of knee replacement, patella button/resurfacing or not, soft tissue procedures outside of standard practise, is collected through patients' medical journals at the 6 week follow up.
Description of post-operative physical therapy management | 6 weeks after surgery; 3 months after surgery; 1 year after surgery
  Brief description of post-operative physical therapy management for all patients is collected via forms at the 6-, 12- and 52-week post-operative follow-up assessments.
Adverse events | From baseline to 1 year after surgery
  Adverse events, such as injuries during intervention participation, re-surgeries, post-operative infections and deaths, are recorded for all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Ljung, PhD-student, Study Director — Linkoeping University
Locations (1):
- Linkoping University, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No
The data that supports the findings of this study will be available on aggregated level from the corresponding author (ML) upon reasonable request after study completion